CLINICAL TRIAL: NCT04799145
Title: Basic Mobility and Balance Performance of Low Active Transfemoral Prosthesis Users With Mobili Knee (a Powered Microprocessor-controlled Knee Prosthesis)
Brief Title: Basic Mobility and Balance Performance of Low Active Transfemoral Prosthesis Users With a Powered Prosthetic Knee
Status: Completed | Type: Interventional
Sponsor: Össur Iceland ehf (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CII2020111613
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-10

CONDITIONS: Prosthesis User; Amputation

STUDY DESIGN:
Intervention Model Description: prospective case series design, within subject comparison
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Investigational device (Experimental): All subjects performed outcome measures on their prescribed knee and the investigational device for comparison.
  Interventions: Device: Investigational device; Device: Prescribed device

INTERVENTIONS:
Device: Investigational device — Motorized microprocessor controlled prosthetic knee.
Device: Prescribed device — Passive microprocessor controlled knee and mechanical knee

SUMMARY:
This was a prospective case series design investigation with 6 prosthesis user subjects. Subjects performed the Timed up and go (TUG) test and the two minute walk test (2MWT) along with some activities of daily living (ADL), on their prescribed knee as well as the investigational device at two separate visits. Performance was compared and statistically analyzed.

DETAILED DESCRIPTION:
Participants were consented, and all tests were conducted at the Össur Motion lab Grjótháls 1-5, 110 Reykjavik.

There were two scheduled study events. At the initial visit, the first study event, for each subject a researcher qualified to obtain informed consent seated the subject and proceeded as described in chapter 13.7 Informed consent in [2].

Prior to fitting the subject was asked to provide feedback on their prescribed prosthesis, by filling in a questionnaire and perform AMPro, LCI (modified), TUG test, 2MWT and other validation activities (stand to sit, sit to stand, level ground, stair and ramp walking), as applicable. The users were fitted within the standard methods of prosthetic fitting, alignment, introduction, training and walking on various terrain.

After initial fitting subjects carried out validation tasks (stand to sit, sit to stand tasks, level ground walking at different speeds, stair and ramp walking), stroop test (cognitive loading) and FSST on the investigational device, after which they answered an in-house questionnaire to provide feedback.

During the second event, subjects were fitted with the investigational device and asked to perform the TUG, 2MWT and any validation tasks that could not be completed at visit 1 on the investigational device due to time restraints or subject condition.

If for some reason all tasks could not be completed at visit 1 and 2 due to time restraints or subject condition, a third visit was added.

Subjects did not wear the device home between visits.

Statistical Considerations:

Outcomes were inspected for normality. If the data was deemed to have a normal distribution the hypothesis was tested using a two-tailed, paired t-test (Only hypothesis A and B). If data was deemed non-normal that hypothesis was tested using a Wilcoxon signed rank test. Significance level (alpha) will be set at 0.05.

Other endpoints and acceptance criteria were assessed with descriptive statistics only.

ELIGIBILITY:
Inclusion Criteria:

* 50Kg< body weight < 116Kg
* Cognitive ability to understand all instructions and questionnaires in the study;
* K1-K2 unilateral transfemoral amputees
* Allows for 37mm knee center height to dome of pyramid alignment
* Age ≥ 18 years
* Willing and able to participate in the study and follow the protocol
* Comfortable and stable socket fit (5 or over on the SFCS)

Exclusion Criteria:

* Users with cognitive impairment
* Users aged <18y
* Bilateral amputees
* Users with stump pain affecting their functional mobility
* Users with socket problems
* Users with co-morbidities in the contra-lateral limb, which significantly affect their functional mobility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All subjects performed outcome measures on their prescribed knee and the Mobili Knee investigational device for comparison.
  Power Knee Mainstream - Balance / Mobili Knee: Motorized microprocessor controlled prosthetic knee.
  Prescribed device: Passive microprocessor controlled knee and mechanical knee
Period: Overall Study
Arm/Group | All Participants
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All subjects performed outcome measures on their prescribed knee and the investigational device for comparison.
  investigational device: Motorized microprocessor controlled prosthetic knee.
  Prescribed device: Passive microprocessor controlled knee and mechanical knee
Arm/Group | All Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Iceland | 6
Ampro [Mean (Standard Deviation); unit: Total Score] — Amputee Mobility Predictor, a test that determines the mobility level of people with amputation. The test subjects receive points for each task depending on their performance. At the end, all points are added up to an overall score. Following scores correspond to the respective activity level: 0-8 (K0); 9-20 (K1); 21-28 (K2); 29-36 (K3); 37-43 (K4). Where users falling in K3 and K4 are considered higher active prosthetic users and users with a K2 level or lower are considered to be lower active prosthetic users.
  Total Score | 33 (6)

OUTCOME MEASURES:

1. Primary Outcome: Timed Up and Go Test (TUG Test)
Description: Subjects are timed while completing a task of getting up from a chair, walking 3 meters at self-selected walking speed, turning around a cone and returning to sit down in the chair.Time is stopped from leaving the chair until the subject is sitting again. The time is measured in seconds. The faster the subject can complete the task the better. Results correlate with gait speed, balance, functional level, the ability to go out, and can follow change over time. It is assumed that subjects that take longer than 14s to complete the TUG might have a higher risk for falls.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | All Participants
Number analyzed (Participants) | 6
seconds
  Prescribed prosthesis | 13.3 (4.9)
  Power Knee | 16.8 (4.5)

2. Secondary Outcome: 2 Minute Walk Test
Description: Subjects walk at self-selected walking speed for 2 minutes, they shall walk as far as possible
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | All Participants
Number analyzed (Participants) | 6
meters
  Prescribed prosthesis | 108.7 (36.7)
  Power Knee | 102.1 (17.9)

ADVERSE EVENTS:
Time Frame: during each study visit while the investigational device was used (half a day), no home use between visits, up to 3 visits per subject over a period of 2 weeks
Arm/Group | Investigational Device
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT04799145/Prot_SAP_001.pdf